CLINICAL TRIAL: NCT03350256
Title: BurstDR™ micrOdosing stimuLation in De-novo Patients
Acronym: BOLD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SJM-CIP-10215
Record Dates: First submitted 2017-11-10; First posted 2017-11-22 (Actual); Results first posted 2020-03-19 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Pain, Intractable; Pain, Back
MeSH Terms: conditions — Pain, Intractable; Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Microdosing group (Experimental): Stimulation will be delivered at with different microdosing setting to identify the optimal parameter values for each patient.
  Interventions: Device: Stimulation will be delivered at with different microdosing setting to identify the optimal parameter values for each patient.

INTERVENTIONS:
Device: Stimulation will be delivered at with different microdosing setting to identify the optimal parameter values for each patient. — BurstDR spinal cord stimulation will be delivered with different ON/OFF periods to identify the best setting for each patients.

SUMMARY:
The purpose of this study is to evaluate the therapeutic efficacy of microdosing BurstDR stimulation in spinal cord stimulation (SCS) patients with chronic intractable back and/or leg pain.

DETAILED DESCRIPTION:
Microdosing BurstDR consists of periods during which stimulation is delivered with standard BurstDR stimulation parameters alternated with periods during which no stimulation is being delivered.

In this study the investigators propose to evaluate therapeutic efficacy of BurstDR microdosing, and determine optimal microdosing programming parameters in chronic pain patients, who are eligible for SCS therapy.

ELIGIBILITY:
Inclusion Criteria:

* Subject is able to provide informed consent to participate in the study;
* Subject diagnosed with chronic intractable pain associated with back and/or limbs;
* Subject is 18 years of age or older;
* Subject has failed to respond to at least 6 months of conventional treatment which may include pharmacological treatment, physical therapy, epidural injections;
* Subject has a back and/or leg pain intensity of at least 6.0 cm out of 10.0 cm on the average back and/or leg pain visual analogue scale at baseline;
* Subject's medical record has been evaluated by the Investigator to ensure that the subject is a good candidate for a neurostimulation system;
* Subject is on stable pain medications with a total opioid for at least 28 days prior to enrolling in this study, and is willing to stay on those medications with no dose increase until the 3 month visit;
* Subject is willing to cooperate with the study requirements including compliance with the regimen and completion of all office visits;
* Female candidates of child-bearing potential agree to commit to the use of an effective method of contraception (including but not limited to sterilization, barrier devices, oral contraceptives, intrauterine devices (IUDs), condoms, rhythm method, or abstinence) for the duration of the study

Exclusion Criteria:

Subject has a current diagnosis of a coagulation disorder, bleeding diathesis, progressive peripheral vascular disease, post-herpetic neuralgia or uncontrolled diabetes mellitus;

* Subject is currently participating in a clinical investigation that includes an active treatment arm;
* Subject has been implanted with or participated in a trial period for a neurostimulation system;
* Subject has an infusion pump;
* Subject has evidence of an active disruptive psychological or psychiatric disorder as determined as per standard of care;
* Subject has a current diagnosis of a progressive neurological disease as determined by the Investigator;
* Subject is immunocompromised;
* Subject has an existing medical condition that is likely to require repetitive MRI evaluation in the future (i.e. epilepsy, stroke, multiple sclerosis, acoustic neuroma, tumor);
* Subject has history of cancer requiring active treatment in the last 12 months;
* Subject has an existing medical condition that is likely to require the use of diathermy in the future;
* Subject has documented history of allergic response to titanium or silicone;
* Subject has a documented history of substance abuse (narcotics, alcohol, etc.) or substance dependency in the 6 months prior to baseline data collection;
* Subject is a female candidates of child bearing potential that are pregnant (confirmed by positive urine/blood pregnancy test);
* Subject has life expectancy of less than 6 months;
* Subject is involved in an injury claim under current litigation

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2019-07-02 (Actual); Study Completion 2019-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy R Deer, MD, Principal Investigator — The Center for Pain Relief
Locations (5):
- United States (5):
  - Thrive Clinic, Santa Rosa, California
  - Nevada advanced pain specialists, Reno, Nevada
  - OnSite Clinical Solutions, Asheville, North Carolina
  - Ambulatory Surgery Center of Killeen, Killeen, Texas
  - Premier Pain Solutions, Charleston, West Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Microdosing Group
Started | 60
Spinal Cord Stimulation Trial | 50 (Subject that underwent SCS trial)
Permanent Implant | 35 (subjects that underwent permanent SCS implant)
1 Month Follow up | 30
3 Month Follow up | 27
6 Month Follow up | 24
Completed | 24
Not Completed | 36
Not completed — Inclusion/exclusion violation | 4
Not completed — Recommended for other therapies | 2
Not completed — Protocol Violation | 3
Not completed — Non compliance | 2
Not completed — Denial by insurance | 1
Not completed — Adverse Event | 2
Not completed — Trial failure | 12
Not completed — Did not proceed to permanent implant | 3
Not completed — Withdrawal by Subject | 3
Not completed — Subject moving out of state | 1
Not completed — Lost to Follow-up | 1
Not completed — Lack of Efficacy | 2

BASELINE CHARACTERISTICS:
Population: Included subjects that started the SCS trial (50). One subjects had missing demographic data
Arm/Group | Microdosing Group
Number analyzed (Participants) | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.8 (3.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 49
duration of pain [Mean (Standard Deviation); unit: years] — Population: One subject had missing data for duration of pain
  years
    number analyzed (Participants) | 48
    (all) | 9.98 (3.31)

OUTCOME MEASURES:

1. Primary Outcome: Change in Visual Analog Scale Pain (VAS) Scores Between Baseline and Trial Stimulation
Description: Pain questionnaire - (Scale is 0-100 mm with 0 meaning no pain and 100 meaning worst pain imaginable)
Time Frame: baseline and 1 week after trial lead implant (trial stimulation)
Population: Change in visual analogue scale score between baseline and spinal cord stimulation (SCS) trial missing data for 3 subjects
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Microdosing Group
Number analyzed (Participants) | 47
units on a scale | -46.28 (23.83)

2. Primary Outcome: Change in Visual Analog Scale Pain Scores Between Baseline and Follow up 1
Description: Pain questionnaire - (Scale is 0-100 mm with 0 meaning no pain and 100 meaning worst pain imaginable)
Time Frame: Baseline and 1 month follow up visit
Population: Change in VAS score between baseline and 1 month follow up missing data for 2 subjects
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Microdosing Group
Number analyzed (Participants) | 28
units on a scale | -41.07 (24.74)

3. Primary Outcome: Change in Visual Analog Scale Pain Scores Between Baseline and Follow up 2
Description: Pain questionnaire - (Scale is 0-100 mm with 0 meaning no pain and 100 meaning worst pain imaginable)
Time Frame: Baseline and 3 month follow up visit
Population: Change in VAS between baseline and 3 month follow up missing data for 2 subject
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Microdosing Group
Number analyzed (Participants) | 25
units on a scale | -36.56 (29.53)

4. Primary Outcome: Change in Visual Analog Scale Pain Scores Between Baseline and Follow up 3
Description: Pain questionnaire - (Scale is 0-100 mm with 0 meaning no pain and 100 meaning worst pain imaginable)
Time Frame: Baseline and 6 month follow up visit
Population: Change in VAS score between baseline and 6 months visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Microdosing Group
Number analyzed (Participants) | 24
units on a scale | -36.62 (29.54)

5. Secondary Outcome: Change in Quality of Life Between Baseline and Trial Stimulation
Description: Questionnaire on quality of life using european quality of life - 5 dimension questionnaire (EQ-5D) - (Scale is between 0 and 1 with 0 being worse quality of life and 1 best quality of life)
Time Frame: Baseline and 1 week after trial lead implant (trial stimulation)
Population: Change in EQ-5D score between baseline and SCS trial
  1 subject had missing data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Microdosing Group
Number analyzed (Participants) | 49
score on a scale | 0.172 (0.1625)

6. Secondary Outcome: Change in Quality of Life Between Baseline and Follow up 1
Description: as for outcome 5
Time Frame: Baseline and 1 month follow up visit
Population: Change in EQ-5D score between baseline and 1 month follow up Two subjects had missing data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Microdosing Group
Number analyzed (Participants) | 28
score on a scale | 0.148 (0.121)

7. Secondary Outcome: Change in Quality of Life Between Baseline and Follow up 2
Description: as for outcome 5
Time Frame: Baseline and 3 month follow up visit
Population: Change in EQ-5D score between baseline and 3 month follow up One subjects had missing data
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Microdosing Group
Number analyzed (Participants) | 26
score on a scale | 0.106 (0.209)

8. Secondary Outcome: Change in Quality of Life Between Baseline and Follow up 3
Description: as for outcome 5
Time Frame: Baseline and 6 month follow up visit
Population: Change in EQ-5D score between baseline and 6 month follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Microdosing Group
Number analyzed (Participants) | 24
score on a scale | 0.148 (0.136)

9. Secondary Outcome: Change in Disability Index Between Baseline and Trial Stimulation
Description: questionnaire on disability, Oswestry Disability Index (ODI) - (Scale is between 0 and 100 with 0 being no disability and 100 worst disability)
Time Frame: Baseline and 1 week after trial lead implant (trial stimulation)
Population: Change in ODI score between baseline and SCS trial 3 subjects had missing data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Microdosing Group
Number analyzed (Participants) | 47
score on a scale | -17.6 (18.15)

10. Secondary Outcome: Change in Disability Index Between Baseline and and Follow up 1
Description: as for outcome 9
Time Frame: Baseline and 1 month follow up visit
Population: Change in ODI score between baseline and 1 month follow up 2 subjects had missing data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Microdosing Group
Number analyzed (Participants) | 28
score on a scale | -12.76 (14.5)

11. Secondary Outcome: Change in Disability Index Between Baseline and and Follow up 2
Description: as for outcome 9
Time Frame: Baseline and 3 month follow up visit
Population: Change in disability score between baseline and 3 month follow up Two subjects had missing data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Microdosing Group
Number analyzed (Participants) | 26
score on a scale | -17 (19.1)

12. Secondary Outcome: Change in Disability Index Between Baseline and and Follow up 3
Description: questionnaire on disability (ODI) - (Scale is between 0 and 100 with 0 being no disability and 100 worst disability)
Time Frame: Baseline and 6 month follow up visit
Population: Change in disability score between baseline and 6 month follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Microdosing Group
Number analyzed (Participants) | 24
score on a scale | -15.5 (16.6)

13. Secondary Outcome: Change in Pain Catastrophizing Scale Between Baseline and Trial Stimulation
Description: Questionnaire on pain catastrophizing, Pain Catastrophising Scale (PCS) - (Scale is between 0 and 52 with 0 being no catastrophising and 52 worst catastrophising)
Time Frame: Baseline and 1 week after trial lead implant (trial stimulation)
Population: Change in PCS between baseline and SCS trial One subject had missing data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Microdosing Group
Number analyzed (Participants) | 49
score on a scale | -8.98 (12.3)

14. Secondary Outcome: Change in Pain Catastrophizing Scale Between Baseline and Follow up 1
Description: as for outcome 13
Time Frame: Baseline and 1 month follow up visit
Population: Change in PCS score between baseline and 1 month follow up 2 subjects had missing data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Microdosing Group
Number analyzed (Participants) | 28
score on a scale | -12.17 (12.83)

15. Secondary Outcome: Change in Pain Catastrophizing Scale Between Baseline and Follow up 2
Description: Questionnaire on pain catastrophizing (PCS) - (Scale is between 0 and 52 with 0 being no catastrophising and 52 worst catastrophising)
Time Frame: Baseline and 3 month follow up visit
Population: Change in PCS between baseline and 3 month follow up 2 subjects had missing data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Microdosing Group
Number analyzed (Participants) | 26
score on a scale | -13.32 (14.38)

16. Secondary Outcome: Change in Pain Catastrophizing Scale Between Baseline and Follow up 3
Description: as for outcome 13
Time Frame: Baseline and 6 month follow up visit
Population: Change in PCS score between baseline and 6 month follow up
  1 subject had missing data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Microdosing Group
Number analyzed (Participants) | 23
score on a scale | -13.42 (12.68)

17. Other Pre Specified Outcome: Stimulation ON/OFF Ratio
Description: Percentage of patients using each ON/OFF ratio
Time Frame: 6 month follow up visit
Measure: Count of Participants; unit: Participants
Arm/Group | Microdosing Group
Number analyzed (Participants) | 24
Participants
  subjects using 360 seconds OFF intervals | 11
  subjects using 240 seconds OFF intervals | 3
  subjects using 150 seconds OFF intervals | 3
  subjects using 120 seconds OFF intervals | 3
  subjects using 90 seconds OFF intervals | 4

ADVERSE EVENTS:
Time Frame: From enrollment to completion of the study at 6 month follow up.
Arm/Group | Microdosing Group
All-Cause Mortality (participants affected / at risk) | 0/60
Serious Adverse Events (participants affected / at risk) | 2/60
Other Adverse Events (participants affected / at risk) | 3/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Microdosing Group (N=60)
Subject fractured <1 vertebrae (compression) and was hospitalized overnight (Injury, poisoning and procedural complications) | 1 (1)
Hospitalization for abdominal pain (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Microdosing Group (N=60)
Trial lead migration (Injury, poisoning and procedural complications) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-19): https://cdn.clinicaltrials.gov/large-docs/56/NCT03350256/Prot_SAP_000.pdf